CLINICAL TRIAL: NCT01780727
Title: Echocardiography-guided Hemodynamic (EGHEM) Management Strategy to Improve Clinical Outcomes for Elderly Patients With Left Ventricular Diastolic Dysfunction (LVDD) Undergoing Non-cardiac Surgery
Brief Title: Echo-guided Hemodynamic Management Strategy in Elderly Patients Undergoing Noncardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0630-12-FB
Record Dates: First submitted 2013-01-23; First posted 2013-01-31 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ventricular Dysfunction, Left; Major Adverse Cardiac Events
Keywords: echocardiography; hemodynamic management
MeSH Terms: conditions — Ventricular Dysfunction, Left; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Arm 1 receives normal saline per the standard of care determined by the anesthesiologist.
  Arm 2 receives normal saline or furosemide per the results of the intraoperative echocardiogram.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Hemodynamic Management (SHEM) (No Intervention): use of standard hemodynamic management
- EGHEM (Experimental): use of echocardiography guided hemodynamic management to control fluid and drug therapy.
  Interventions: Procedure: EGHEM

INTERVENTIONS:
Procedure: EGHEM — Echocardiography guided hemodynamic management. Subjects in this arm will undergo intraoperative transesophageal echocardiography as part of the study.
  Arms: EGHEM

SUMMARY:
Elderly patients are the fastest growing surgical population and have an increased risk of postoperative cardiac problems. Diastolic dysfunction, or the reduced ability of the heart' s ventricles to fill completely, is common in the elderly population and increases the risk of major adverse cardiac events after surgery. This study will measure diastolic filling and implement fluid and drug management during surgery to determine whether this reduces serious cardiac events related to diastolic dysfunction after surgery in this high-risk population.

DETAILED DESCRIPTION:
Elderly patients are the fastest growing surgical population and present with increased risk of postoperative cardiac problems, especially congestive heart failure. Diastolic dysfunction is common in the elderly population and increases the risk of major adverse cardiac events after surgery. This project will use dynamic measurements of diastolic filling pressures by echocardiography for goal-directed fluid and drug management during surgery to determine whether this reduces serious cardiac events related to diastolic dysfunction after surgery in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older
* Echocardiographic Evidence of Grade I, II or III LVDD on Preoperative Transthoracic Echocardiography (TTE) examination
* Undergoing Vascular Surgery including but not limited to : Lower extremity bypass,Open abdominal aortic aneurysm repair

Exclusion Criteria:

* Patients with expected hospital stay < 24 hours
* Inability to undergo TEE and Transesophageal Echocardiography(TTE)
* Clinical evidence/suspicion of elevated Intercranial Pressure (ICP)
* Preoperative shock or systemic sepsis
* Emergency operation
* American Society of Anesthesiologists Status V
* Participation in another clinical trial
* General Anesthesia not planned for procedure

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Patients who undergo dynamic heart function changes during surgery | 2 years
  We will test the hypothesis that Left Ventricular Diastolic Dysfunction (LVDD) undergoes dynamic changes perioperatively.
  A. We will preoperatively identify 200 elderly subjects to provide 80% power to detect a change in LVDD undergoing noncardiac surgery using a 0.01 level two-sided paired t-test.
  B. We will assess changes in LVDD in these subjects based on hourly intraoperative echocardiography data points.

SECONDARY OUTCOMES:
Safety of Echo-Guided Hemodynamic Management during surgery | 1 year
  We will test the hypothesis that goal-directed Echocardiography Guided Hemodynamic Management (EGHEM) used in elderly subjects with LVDD improves postoperative clinical outcomes.
  A. We will determine the ability of goal-directed EGHEM to maintain or improve intraoperative LVDD.
  B. We will determine the ability of goal-directed EGHEM to reduce postoperative Major Adverse Cardiac Event (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Sasha K Shillcutt, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States